CLINICAL TRIAL: NCT05722548
Title: Efficacy of Rectal Indomethacin in Prevention of Post-pancreatectomy Acute Pancreatitis-A Randomized Controlled Trial
Brief Title: Efficacy of Rectal Indomethacin in Prevention of Post-pancreatectomy Acute Pancreatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yingbin Liu, MD, PhD, FACS, prof., Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LYBWWG2023
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Pancreatectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients will be administered 100mg of Indomethacin Suppository sigle dose at the time of induction of anesthesia with Standard Medical Treatment
  Interventions: Drug: Indomethacin suppository; Other: Standard Medical Treatment
- Group B (Active Comparator): Standard Medical Treatment
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Drug: Indomethacin suppository — 100mg of Indomethacin Suppository sigle dose at the time of induction of anesthesia
  Arms: Group A
Other: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy of rectal indomethacin in prevention of post-pancreatectomy acute pancreatitis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of rectal indomethacin in prevention of post-pancreatectomy acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

*All patients planned to undergo pancreatectomy.

Exclusion Criteria:

* asthma
* allergic reactions to NSAIDs
* CKD
* internal hemorrhoids
* anti-platelet medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Post-pancreatectomy Acute Pancreatitis | 2 weeks after pancreatectomy

SECONDARY OUTCOMES:
Pancreatic Fistula | 30 days after pancreatectomy
Peripancreatic abscess | 30 days after pancreatectomy
Length of hospital stay | 30 days after pancreatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Yingbin Liu, PHD, Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No